CLINICAL TRIAL: NCT06829563
Title: A Phase Ia/Ib, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose/Multiple Dose Study of RZ-629 to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect in Healthy Subjects and T2D Patients.
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RZ-629 in Healthy Subjects and T2D
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rezubio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RZ-629-EN-01
Record Dates: First submitted 2025-01-22; First posted 2025-02-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants, the investigator, the clinic personnel, the bioanalytical laboratory staff, and other study-related personnel will remain blinded to all randomization assignments. Selected individuals not involved in conducting this trial, including Institutional Review Board (IRB) members, may have access to the unblinded data as needed for safety or other data review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1 - RZ-629 (Experimental): Part 1 - SAD cohorts: participants receiving RZ-629
  Interventions: Drug: RZ-629
- Part 1 - Placebo (Placebo Comparator): Part 1 - SAD cohorts: participants receiving matching placebo
  Interventions: Drug: Placebo
- Part 2 - Food effect (fasted) (Experimental): Part 2 - PK profile of RZ-629 in fasted condition
  Interventions: Drug: RZ-629; Other: Fasted
- Part 2 - Food effect (fed) (Experimental): Part 2 - PK profile of RZ-629 in fed condition
  Interventions: Drug: RZ-629; Other: Fed
- Part 3 - MAD placebo (Placebo Comparator): Part 3 - MAD matching placebo
  Interventions: Drug: Placebo
- Part 3 - MAD RZ-629 (Experimental): Part 3 - multiple doses of RZ-629 in healthy participants
  Interventions: Drug: RZ-629
- Part 3 - MAD placebo in T2D (Placebo Comparator): Part 3 - Multiple doses of matching placebo in T2D
  Interventions: Drug: Placebo
- Part 3 - MAD RZ-629 in T2D (Experimental): Part 3 - Multiple doses of RZ-629 in T2D
  Interventions: Drug: RZ-629

INTERVENTIONS:
Drug: RZ-629 — Administered orally
  Arms: Part 1 - RZ-629; Part 2 - Food effect (fasted); Part 2 - Food effect (fed); Part 3 - MAD RZ-629; Part 3 - MAD RZ-629 in T2D
Drug: Placebo — Administered orally
  Arms: Part 1 - Placebo; Part 3 - MAD placebo; Part 3 - MAD placebo in T2D
Other: Fasted — Participants will be treated with RZ-629 in fasted or fed condition and then cross over after washout
  Arms: Part 2 - Food effect (fasted)
Other: Fed — Participants will be treated with RZ-629 in fasted or fed condition and then cross over after washout
  Arms: Part 2 - Food effect (fed)

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) biomarkers in single ascending doses (SAD), food effect, and multiple doses studies of RZ-629 in healthy participants and T2D.

DETAILED DESCRIPTION:
This study comprises of 3 parts - Part 1, Part 2, and Part 3.

Part 1 (SAD in healthy participants) - A total of 50 healthy subjects will be allocated to 5 groups in the SAD study. Each group includes 10 subjects (8 subjects will receive RZ-629 and 2 receive placebo). All subjects will check-in on the day before the administration (Day -1) and on Day 1. Each subject in fasted state will be randomly assigned to receive a single oral dose of RZ-629 or placebo. Subjects will remain in the clinical research unit (CRU) through the completion of the safety/tolerability evaluation. The safety review committee (SRC) will review all safety data and blinded summary of available PK data through the safety follow-up and decide to proceed to the next dose level.

Part 2 (food effect in healthy participants) - A total of 12 healthy subjects will be enrolled to FE study. Subjects in the FE group will be divided into subgroup A and subgroup B equally. During period 1, subjects in subgroup A will receive a single oral dose of RZ-629 tablet with 240 mL of water following a fast of at least 10 hours. Water is not allowed 1 h predose until 1 h post dose. Food or drinks are not allowed until 4 h after the dosing. Subjects in subgroup B will received the dose of RZ-629 tablet with 240 mL of water following a standardized high-calorie meal consumed after an overnight fast of at least 10 h. The meal is approximately 500 kcal, composed of approximately 50% carbohydrates, 30% fat, and 20% protein.The high-fat meal should be consumed within 30 minutes. The 25 mg RZ-629 tablet should be administrated 30 minutes after starting the high-calorie meal. Water is not allowed 1 h predose until 1 h post dose. No food or drinks are allowed for 4 hours post-dose for all subjects in subgroup B.

During period 2, administration will be performed in a crossover manner, i.e., subjects in subgroup A will receive the study drug after consuming a high-fat meal, and subjects in subgroup B will receive the study drug under fasting conditions. There is a washout period of 10 days between each dose. Relevant PK and PD sampling, and safety assessments will be completed during the study.

Part 3 (multiple doses in healthy subjects and in T2D patients) - A total of 72 subjects will be recruited with each cohort including 8 subjects for multiple doses in healthy subjects (body mass index [BMI] between 19 and 32 kg/m2, 6 on RZ-629 and 2 on placebo) and 12 subjects for multiple doses in T2D patients (BMI between 25 and 40 kg/m2, 9 on RZ-629 and 3 on placebo). Subjects will check in on Day -2 to Day -1 for healthy subjects and Day -2 for T2DM patients after 28 days of screening.

On Day 1, healthy subjects will be randomly assigned to orally receive the RZ-629 or placebo once daily for a consecutive 7 days. After being evaluated by the investigator, patients will leave the CRU on Day 2 and return to the CRU on Day 5, Day 6, Day 7 and stay until Day 10, for safety and tolerability assessments, and will be discharged with the consent of the investigator. All subjects will return to the CRU for safety follow-up on Day 15 + 2.

T2D patients cohorts will be enrolled after safety assessment of multiple doses study in healthy subjects. T2D patients will be randomly assigned to orally receive RZ-629 or placebo once daily for a consecutive 28 days. After being evaluated by the investigator, patients will leave the CRU on Day 2 and return to the CRU on Day 8, Day 15, and Day 22 for biosample collection and safety examination. They will then return to the CRU on Day 27 and stay until the end of Day 29. All subjects will return to the CRU for safety follow-up on Day 35 + 2.

ELIGIBILITY:
Inclusion Criteria: 1. Sign the informed consent form (ICF) before the study, and fully understand the content, process and possible adverse reactions of the trial.

2. Healthy male or female subjects between the ages of 18 and 65 years, inclusive.

3. For part 1, part 2 and part 3 in healthy participants, minimum body weight is 50 kg for males, and 45 kg for females, have a BMI of 18 to 32 kg/m2, inclusive. For part 3 in T2D, BMI is between 25 to 40 kg/m2, inclusive.

4. For part 1, part 2, and part 3 in healthy participants, fasting plasma glucose is between 3.9 mmol/L (70.2 mg/dL) and 6.1 mmol/L (109.8 mg/dL) at screening. For part 3 in T2D, glycosylated hemoglobin A1c (HbA1c) is between 6.5% and 10.5%, inclusive, and FPG ≤ 13.3 mmol/L at screening.

5. For part 1, part 2, and part 3 in healthy participants, participants are in good health, with no clinically relevant acute or chronic medical conditions or severe diseases of the cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, respiratory, blood, immune or dermatological systems, as judged by the investigator. For part 3 in T2D, participants are diagnosed with T2DM for more than 1 year, and on a stable dose of dipeptidyl peptidase IV inhibitor (DPP-4i) monotherapy or DPP-4i + Metformin as their only anti-hyperglycemic treatment for at least 3 months prior to the screening visit.

6. With no clinically significant findings from vital signs measurements, physical examination, clinical laboratory evaluations and 12-lead ECG, as judged by the investigator.

7. Subjects must be willing to understand and comply with all research procedures and restrictions and be able to communicate effectively with researchers.

Exclusion Criteria: 1. With a specific history of allergies or known to have multiple allergies.

2. Have experienced acute illnesses within 2 weeks prior to the first dose or are taking concomitant medications.

3. With a history or current presence of dysphagia or diseases that may potentially interfere with drug absorption or metabolism.

4. Subjects and their first-degree relatives with a history of diabetes before screening.

5. With a history of hypoglycemia or with impaired awareness or cognition of hypoglycemic symptoms within 3 months prior to screening.

6. History of previous corrected QT interval (QTc) prolongation or clinically abnormal electrocardiogram (ECG) finding during screening.

7. Have undergone major surgery within the past 6 months, or those planning to undergo surgery during the study period.

8. Have used any medications and dietary supplements within 2 weeks prior to the first dose.

9. Within 48 h prior to the first dose, have consumed food or beverages containing caffeine, alcohol, or concentrated tea, or those who have consumed special diets and/or purine-rich diets or have other factors that may affect drug absorption, distribution, metabolism, or excretion.

10. Have received vaccinations within 4 weeks prior to the first dose or plan to receive vaccinations during the trial.

11. Have participated in other clinical trials within 3 months prior to the first dose, or those planning to participate in other trials during the study period.

12. Have donated blood and blood products (including plasma) within 3 months prior to the first dose or have experienced non-physiological blood loss of ≥ 400 mL within 6 months.

13. Have consumed an average of more than 14 units of alcohol per week within the past 12 months prior to screening.

14. Have smoked more than 5 cigarettes per day within the past 3 months or cannot stop using any tobacco products during the study.

15. With a history of drug abuse within the past 12 months or positive drug abuse at screening.

16. With positive results for serology of infectious diseases at screening. 17. Cannot tolerate venipuncture/indwelling needle or have a history of vasovagal syncope.

18. Subjects deemed unsuitable for participation in this trial by the investigator due to other factors.

19. With chronic or acute gastrointestinal inflammation. 20. Abnormal liver function tests: ALT or AST > 2×ULN, or TBIL > 1.5×ULN. 21. Use of drugs that may affect glucose metabolism (e.g., systemic steroids, nonselective β-blockers, monoamine oxidase inhibitors) within 1 month prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting 1 or more treatment-emergent adverse events | Baseline to day 7
  Safety assessment of RZ-629 treatment evaluated by proportion of participants with adverse events, laboratory tests, vital signs, and ECGs.

SECONDARY OUTCOMES:
Area under the concentration-time curve [AUC] of plasma RZ-629 | Baseline to day 7
  Collect blood samples to evaluate AUC
Maximum concentration [Cmax] of plasma RZ-629 | Baseline to Day 7
  Collect blood samples to evaluate Cmax
Changes from baseline in insulin and incretins | Baseline to Day 7
  Collect blood samples to evaluate changes from baseline in insulin and incretins
Changes in metabolic parameters in multiple doses study in T2D | Day 1 to week 4
  Changes from baseline in body weight, blood glucose, HbA1c, and lipid profile in multiple doses study in T2D

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No